CLINICAL TRIAL: NCT03982550
Title: Cerebrovascular Mechanisms of Cognitive Enhancement After Periodized Resistance Training in Older Adults
Brief Title: Resistance Training and Neuroimaging
Acronym: RTNI
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Todd Schroeder (Other)
Collaborators: Southern California Clinical and Translational Science Institute (Unknown)
Responsible Party: Sponsor-Investigator, Todd Schroeder, Associate Professor of Clinical Physical Therapy, University of Southern California
Organization: University of Southern California (Other)
Allocation: Non-Randomized | Model: Crossover | Masking: None | Purpose: Basic Science
Other Study IDs: HS-17-00770
Record Dates: First submitted 2019-06-05; First posted 2019-06-11 (Actual); Last update posted 2022-05-20 (Actual); Status verified 2022-05

CONDITIONS: Cognitive Decline; Cerebrovascular Function
MeSH Terms: conditions — Cognitive Dysfunction

STUDY DESIGN:
Intervention Model Description: There are two phases in this single-group study: an initial control period and an intervention period. All control periods will take place before the RT intervention to ensure that results are not confounded by detraining effects or long-term cognitive benefits of RT.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control Period (No Intervention): Participants will serve as their own controls. All 12-week control periods will take place before the RT intervention to ensure that results are not confounded by detraining effects or long-term cognitive benefits of RT. In addition, a control period equal in duration to the intervention allows direct within-subjects statistical comparisons, accounting for each participants' baseline and rate of aging - i.e. age-associated cognitive decline and arterial stiffening. Participants will not be monitored, but may be contacted for scheduling.
- Intervention Period (Experimental): Participants will perform a periodized and progressive total-body RT program emphasizing development of lower and upper body strength. All 36 training sessions (3 days per week for 12 weeks) will be performed at the CERC, supervised by an exercise specialist. Participants will be encouraged to continue normal activities of daily living and eating routines outside the RT program of the present study. Because this is a proof-of concept study on normal aging, participants may be contacted for scheduling, but will not be monitored outside of training.
  Interventions: Behavioral: Periodized Resistance Training

INTERVENTIONS:
Behavioral: Periodized Resistance Training — Mesocycle I (weeks 1-4) will emphasize muscular hypertrophy to develop a muscular and metabolic base for more intense training in later phases. Training bouts will consist of 4-6 resistance exercises with 2-4 sets per exercise and 8-10 repetitions per set. Mesocycles II (weeks 5-8) and III (weeks 9-12) will emphasize strength development. Training bouts will consist of 4-6 resistance exercises with 3-5 sets per exercise, 4-6 repetitions per set, and linear increases in intensity over time. These parameters were chosen to maximize performance on 4-6 repetition maximum (RM) testing post-intervention, according to the principle of specificity - i.e. specific adaptation to imposed demands.The training loads used will be individually progressed in a safe and effective manner, in order to employ a progressive overload/challenge to the neuromuscular system and elicit the greatest training-induced neuromuscular adaptations possible.
  Arms: Intervention Period

SUMMARY:
Aging tends to compromise the ability to solve problems, remember details, and process information. At the extreme level, this normal cognitive decline can interfere with independent living. Because most brain dysfunctions become irreversible before patients show clear signs in the clinic, there is a pressing need to prioritize preventative countermeasures. Exercise is a promising strategy to slow or reverse these losses. While most studies have looked at running or cycling exercise, little is known about the effects of weight lifting exercise. In addition, vascular health is intimately linked with cognitive abilities and risk of stroke, making it a primary target for intervention. Previous weight lifting studies suggest that blood vessels in the brain are a likely site of adaptation.

The goal of this research is to understand how weight lifting exercise improves cognitive function in older adults. Specifically, the contribution of blood vessel changes in the brain after 12 weeks of weight lifting exercise 3 days per week. These vascular improvements may provide the link between physical and cognitive health, while simultaneously reducing the risk of cardiovascular disease and stroke. To determine this, advanced brain imaging techniques will be used to measure blood flow/volume changes in the brain non-invasively. Physical capacity (i.e. strength), body composition (i.e. lean mass, fat mass), and blood markers will also be assessed using standard protocols, and each of these variables will be tested for their relationship with cognitive functions.

Understanding how weight lifting exercise improves cognitive function will support the development of comprehensive treatments targeting overall brain health. With no current cures for dementia, this information will be vital in prescribing exercise for specific patient needs to reducing the risk of dementia and stroke. In addition, the promise of exercise therapies extends beyond the target disease, having further benefits to the well-being of participants. These types of treatments positively impact fundamental aging processes, and thus reduce the risk of all-cause mortality. Even with moderate benefits to a specific disease like dementia, the global impact on healthcare would be substantial.

DETAILED DESCRIPTION:
Exercise is a promising strategy to slow or prevent the progression of cognitive decline and dementia. While resistance training (RT) is a popular form of exercise recommended for older adults for its putative role in the protection against sarcopenia, its effects on brain health have been less-well studied. Previous RT studies involving traditional protocols highlight robust and lasting benefits to fluid cognition. In contrast, little is known about the effects of high-intensity RT with advanced periodization techniques. Such protocols may produce similar improvements in shorter durations, thus improving clinical utility. In addition, the mechanisms of RT-induced cognitive enhancement are not well understood. Defining the dominant neural and physiological processes that underlie these protective effects is essential to explain the variance in cognitive responses and to design optimal treatment strategies for the aging population.

The effectiveness of RT interventions for cognitive health likely depends on maximizing gains in muscular strength. Therefore, the investigators will apply strength and conditioning principles and advanced neuroimaging techniques to a 12-week periodized RT intervention to determine neuroprotective contributions. Cerebrovascular (CV) function is a major component of brain health and a primary mechanism of cognitive enhancement after aerobic training. However, the potential for RT to influence these pathways has not been determined. This study will test and extend previous cross-sectional evidence linking RT with CV function. In addition, RT interventions have been demonstrated to improve systemic vascular function and cognition independently. Thus, the investigators hypothesize that RT improves cognitive function through muscular strength and CV adaptations. The overall goal of this proposal is to investigate changes in cognition and CV function in 23 healthy older adults 60-80 years of age, serving as their own controls, and explore the mechanisms that mediate these effects. To address this goal, the investigators propose the following aims:

Aim 1: To determine whether 12 weeks of periodized RT improves fluid cognition in older adults. The NIH Toolbox® Cognition Battery will be administered to assess changes in executive function, attention, episodic memory, processing speed, working memory, and language. Composite scores will be computed for fluid, crystallized, and global cognitive function.

Hypothesis: A 12-week periodized RT program designed specifically to maximize strength gains improves fluid cognition in healthy older adults.

Aim 2: To evaluate the effects of periodized RT on CV function in older adults. Arterial spin labeling (ASL) MRI techniques will be used to assess changes in CV function by quantifying the effects on resting cerebral blood flow, intracranial vascular compliance, and arterial transit time. Mediation analyses will be performed to determine the mediating effects of CV function on cognition.

Hypothesis: High-intensity RT can improve CV function in healthy older adults.

Aim 3: To explore associations between brain adaptations and potential mechanisms of benefit, including: 1) physical capacity (e.g. muscular strength), body composition, and functional mobility; 2) putative blood markers of exercise-induced brain plasticity; 3) cardiovascular risk factors; and 4) brain morphometry and resting state brain activity. Significant changes will be analyzed for mediation of cognitive function to identify the major pathways that underlie the protective effects of RT.

For the practicality of this study, participants will serve as their own controls. All control periods will take place before the RT intervention to ensure that results are not confounded by detraining effects or long-term cognitive benefits of RT. All participants will undergo testing at baseline, pre-intervention, and post-intervention. The NIH Toolbox Cognition Battery will provide a standard set of comprehensive assessment tools. Three test versions will be used to reduce practice effects. During MRI scans, ASL techniques will be used to assess CV function and standard sequences will be used for structural MRI (e.g. T2-weighted FLAIR and T1-weighted MP-RAGE), resting state function MRI (rfMRI), and diffusion tensor imaging (DTI). Physical outcomes will be assessed using standard testing procedures in exercise physiology research, including blood pressure, body composition, physical function, muscle strength and estimated VO2max. Validated questionnaires for quality-of-life, physical activity, sleep quality, and interpersonal support will be administered.

Participants will perform a periodized and progressive total-body resistance training program emphasizing development of lower and upper body strength. All 36 training sessions (3 days per week for 12 weeks) will be performed at the CERC, supervised by an exercise specialist. Mesocycle I (weeks 1-4) will emphasize muscular hypertrophy to develop a muscular and metabolic base for more intense training in later phases. Training bouts will consist of 4-6 resistance exercises with 2-4 sets per exercise and 8-10 repetitions per set. Mesocycles II (weeks 5-8) and III (weeks 9-12) will emphasize strength development. Training bouts will consist of 4-6 resistance exercises with 3-5 sets per exercise, 4-6 repetitions per set, and linear increases in intensity over time. As in similar RT studies, the training loads used will be individually progressed in a safe and effective manner in order to employ a progressive overload/challenge to the neuromuscular system and elicit the greatest training-induced neuromuscular adaptations possible.

ELIGIBILITY:
Inclusion Criteria:

* Community-dwelling and living independently (without need of assistance).
* Interest and availability for participation in a 12-week planned RT program at the CERC, including pre- and post- testing.
* Competency in English sufficient for assessment and training.
* Able to see and hear sufficiently to participate in RT.
* Not engaged in any structured exercise training outside of this intervention.
* Eligible to undergo MRI.
* Answer NO to all questions on the Physical Activity Readiness Questionnaire (PAR-Q) or receive medical clearance from a physician.

Exclusion Criteria:

* Possible Dementia (score less than or equal to 23 on MMSE).
* History of known neurological disease (e.g. Epilepsy, Multiple sclerosis, Parkinson disease, Alzheimer's disease), cerebral infarct (e.g. Stroke), or traumatic brain injury.
* History of known cardiovascular or metabolic disease or chronic illness which may compromise the patient's ability to safely perform the RT program (e.g. coronary artery disease, arrhythmia, asthma requiring an inhaler during exercise), or presently uncontrolled hypertension (SBP > 140 mmHg or DBP > 90 mmHg). Patient may be required to provide clearance from a physician at the study team's discretion.
* Type 1 or Type 2 Diabetes.
* Changes in chronic pharmacological treatment (e.g. Aspirin, Statins, or ACE inhibitors) or hormone therapy during the intervention period.
* Current treatment for congestive heart failure, angina, uncontrolled arrhythmia, DVT or other cardiovascular event.
* Myocardial infarction, coronary artery bypass grafting, angioplasty or other cardiac condition in the past year.
* Contraindications against MRI (e.g. metal implants, claustrophobia).
* Self-report regular heavy RT in the past 6 months (i.e. "strengthening exercises or lifting weights heavy enough that you could not perform more than 15 repetitions in one set").
* Musculoskeletal injuries interfering with the ability to perform RT or medical conditions for which exercise in contraindicated.

Ages: 60 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2018-07-17 (Actual); Primary Completion 2020-05-16 (Actual); Study Completion 2020-05-16 (Actual)

PRIMARY OUTCOMES:
Change in Fluid Cognition Composite Score | Baseline, after the initial 12-week control period, and after the 12-week intervention period.
  NIH Toolbox Cognition Battery
Change in Cerebral Blood Flow | Baseline, after the initial 12-week control period, and after the 12-week intervention period.
  Arterial Spin Labeling Magnetic Resonance Imaging
Change in Vascular Compliance | Baseline, after the initial 12-week control period, and after the 12-week intervention period.
  Arterial Spin Labeling Magnetic Resonance Imaging
Change in Arterial Transit Time | Baseline, after the initial 12-week control period, and after the 12-week intervention period.
  Arterial Spin Labeling Magnetic Resonance Imaging

SECONDARY OUTCOMES:
Change in Crystallized Cognition Composite Score | Baseline, after the initial 12-week control period, and after the 12-week intervention period.
  NIH Toolbox Cognition Battery
Change in Total Body Strength | Baseline, after the initial 12-week control period, and after the 12-week intervention period.
  Calculated 1-repetition maximum
Change in Body Weight | Baseline, after the initial 12-week control period, and after the 12-week intervention period.
  InBody
Change in Body Fat Percentage | Baseline, after the initial 12-week control period, and after the 12-week intervention period.
  Dual-energy X-Ray Absorptiometry
Change in Lower Extremity Power | Baseline, after the initial 12-week control period, and after the 12-week intervention period.
  Margaria Stair Climb
Change in Systolic Blood Pressure | Baseline, after the initial 12-week control period, and after the 12-week intervention period.
  Cadiovascular Risk Factors
Change in Diastolic Blood Pressure | Baseline, after the initial 12-week control period, and after the 12-week intervention period.
  Cadiovascular Risk Factors
Change in Heart Rate | Baseline, after the initial 12-week control period, and after the 12-week intervention period.
  Cadiovascular Risk Factors
Change in Timed-Up-and-Go | Baseline, after the initial 12-week control period, and after the 12-week intervention period.
  Functional Mobility
Change in Gait Speed | Baseline, after the initial 12-week control period, and after the 12-week intervention period.
  Functional Mobility
Change in Y-Balance Total Score | Baseline, after the initial 12-week control period, and after the 12-week intervention period.
  Functional Mobility
Change in Hippocampal Volume | Baseline, after the initial 12-week control period, and after the 12-week intervention period.
  T1-weighted MP-RAGE
Change in White Matter Lesion Volume | Baseline, after the initial 12-week control period, and after the 12-week intervention period.
  T2-weighted FLAIR

CONTACTS AND LOCATIONS:
Locations (1):
- Clinical Exercise Research Center, Los Angeles, California, United States

IPD SHARING:
Plan to Share IPD: Undecided